CLINICAL TRIAL: NCT01413633
Title: A Novel Technique For Gall Bladder Fundus Retraction In Single Incision Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, MOHAMED ABDELLATIF, md, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: how to do it
Record Dates: First submitted 2011-08-08; First posted 2011-08-10 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Gallbladder Diseases
MeSH Terms: conditions — Gallbladder Diseases | interventions — Cholecystectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cholecystectomy (Experimental): single incision laparoscopic cholecystectomy
  Interventions: Procedure: cholecystectomy

INTERVENTIONS:
Procedure: cholecystectomy — single incision laparoscopic cholecystectomy
  Other Names: SILC

SUMMARY:
The investigators describe a novel technique for GB fundus retraction.

DETAILED DESCRIPTION:
few methods are available for gall bladder (GB) retraction in SILC to replace the usage of ancillary ports imitating retraction from conventional technique, e.g. trans-parietal stitches mini-loop retractor , a Kirschner wire . This technical note describes a novel way to retract the gall bladder fundus.

ELIGIBILITY:
Inclusion Criteria:

* all cases underwent single incision cholecystectomy

Exclusion Criteria:

* none

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
operative time | about 3 hours
  the time from starting the procedure till the skin closure

CONTACTS AND LOCATIONS:
Overall Officials: DRAMADAN ELLITHY, M, Study Chair — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt